CLINICAL TRIAL: NCT02148016
Title: Corneal Epithelium Repair and Therapy Using Autologous Limbal Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, MD, PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013SKL005
Record Dates: First submitted 2014-05-19; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Corneal Disease; Pterygium; Myopia; Hyperopia
Keywords: Corneal disorders; Chemical injury; Pterygium; Refractive error; Myopia; Hyperopia; Cornea; Monocular; Transparent; Transplantation; Visual function
MeSH Terms: conditions — Corneal Diseases; Pterygium; Myopia; Hyperopia; Refractive Errors | interventions — Levofloxacin; Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LSCs and amniotic membrane (Modified Technique) (Experimental): Limbal stem cells (LSCs) from the contralateral eye will be harvested and expanded in feeder-free, chemically defined media for one week on a collagen-coated contact lens. The LSCs on contact lens will be transplanted onto a corneal surface in vivo, following removal of scar tissue due to chemical injury or pterygium. The contact lens will then be covered with amniotic membrane to secure it in place.
  The eye will be treated with antibiotics (levofloxacin) and steroids (betamethasone), and then patched.
  Interventions: Procedure: LSCs and amniotic membrane (Modified Technique); Drug: Levofloxacin; Drug: Betamethasone
- Amniotic membrane only (Traditional Technique) (Active Comparator): Amniotic membrane alone will be used to cover the corneal surface, after removal of scar tissue from a chemical injury or pterygium.
  Interventions: Procedure: Amniotic membrane only (Traditional Technique)
- PRK, LSCs, and amniotic membrane (Modified Technique) (Experimental): Limbal stem cells (LSCs) from the contralateral eye will be harvested and expanded in feeder-free, chemically defined media for one week on a collagen-coated contact lens. The LSCs on contact lens will be transplanted onto a corneal surface in vivo, following photo-refractive keratectomy (PRK). The contact lens will then be covered with amniotic membrane to secure it in place.
  The eye will be treated with antibiotics (levofloxacin) and steroids (betamethasone), and then patched.
  Interventions: Procedure: PRK, LSCs, and amniotic membrane (Modified Technique); Drug: Levofloxacin; Drug: Betamethasone; Drug: Limbal stem cells (LSCs)
- PRK only (Traditional Technique) (Active Comparator): PRK alone will be performed.
  Interventions: Procedure: PRK only (Traditional Technique)

INTERVENTIONS:
Procedure: LSCs and amniotic membrane (Modified Technique) — Limbal stem cells (LSCs) from the contralateral eye will be harvested and expanded in feeder-free, chemically defined media for one week on a collagen-coated contact lens. The LSCs on contact lens will be transplanted onto a corneal surface in vivo, following removal of scar tissue due to chemical injury or pterygium. The contact lens will then be covered with amniotic membrane to secure it in place.
  The eye will be treated with antibiotics (levofloxacin) and steroids (betamethasone), and then patched.
  Arms: LSCs and amniotic membrane (Modified Technique)
Procedure: Amniotic membrane only (Traditional Technique) — Amniotic membrane alone will be used to cover the corneal surface, after removal of scar tissue from a chemical injury or pterygium.
  Arms: Amniotic membrane only (Traditional Technique)
Procedure: PRK, LSCs, and amniotic membrane (Modified Technique) — Limbal stem cells (LSCs) from the contralateral eye will be harvested and expanded in feeder-free, chemically defined media for one week on a collagen-coated contact lens. The LSCs on contact lens will be transplanted onto a corneal surface in vivo, following photo-refractive keratectomy (PRK). The contact lens will then be covered with amniotic membrane to secure it in place.
  The eye will be treated with antibiotics (levofloxacin) and steroids (betamethasone), and then patched.
  Arms: PRK, LSCs, and amniotic membrane (Modified Technique)
Procedure: PRK only (Traditional Technique) — PRK alone will be performed.
  Arms: PRK only (Traditional Technique)
Drug: Levofloxacin
  Arms: LSCs and amniotic membrane (Modified Technique); PRK, LSCs, and amniotic membrane (Modified Technique)
Drug: Betamethasone
  Arms: LSCs and amniotic membrane (Modified Technique); PRK, LSCs, and amniotic membrane (Modified Technique)
Drug: Limbal stem cells (LSCs)
  Arms: PRK, LSCs, and amniotic membrane (Modified Technique)

SUMMARY:
Corneal disease is a leading cause of blindness in the world. A shortage of corneal donor tissue has prevented many patients from regaining vision. Additionally, refractive error such as myopia is a major cause of impaired visual function worldwide. Although refractive error is correctable by procedures that modify the refractive power of the cornea, these procedures often weaken corneal integrity and have risk of complications. This study aims to evaluate the safety and efficacy of corneal surface epithelium repair and regeneration in the treatment of corneal surface diseases and refractive error using autologous limbal stem cell transplantation.

DETAILED DESCRIPTION:
The corneal surface is comprised of a unique type of non-keratinized epithelial cell. These cells are arranged in an orderly fashion, which is essential for vision by maintaining the transparency of the visual axis.

Chemical injury and pterygia may damage the limbus, the zone between the cornea and the bulbar conjunctiva, and cause limbal stem cell (LSC) deficiency. They represent major treatable causes of vision loss worldwide. A shortage of corneal donor tissue prevents many patients from regaining vision, necessitating new treatment strategies to circumvent this limitation. Transplantation of stem cells represents an appealing therapeutic strategy in regenerative medicine, and the use of endogenous stem cells provides a possible solution to the problem of immune rejection.

Currently, LASIK (laser-assisted in situ keratomileusis) is the most commonly performed laser vision correction procedure in the world (over 10 million surgeries each year); however, it has a major disadvantage in that it weakens corneal integrity and structure and predisposes to complications such as keratectasia or keratoconus (bulging of the cornea) and vision loss. An alternative is photo-refractive keratectomy (PRK), which removes the corneal epithelium and anterior stroma while minimizing the incidence of keratectasia or keratoconus. The primary drawbacks of PRK are that it requires a longer recovery time (the corneal epithelium must regenerate from the patient's own LSCs) and may result in blurry vision and pain due to corneal pain nerve fiber exposure after removal of the epithelium. Coverage of exposed corneal stroma tissue immediately after surgery with LSC-derived corneal epithelial cells will solve this key bottleneck and make laser eye surgery safer and more comfortable for millions of people.

It is known that corneal renewal and repair are mediated by stem cells in the limbus. Autologous LSC transplantation has been reported previously (Rama et al.). However, mouse feeder cells were required to expand LSCs in culture. We have successfully developed a feeder-free, chemically defined medium in which to expand LSCs. These expanded LSCs can repair and regenerate corneal surfaces (Ouyang et al., in press).

Hypothesis: The trial will demonstrate whether a new technique, transplantation of LSCs expanded from limbal tissue of the uninjured eye, can improve the visual function of patients with unilateral corneal ocular surface disease. In addition, it will show whether there is more rapid recovery and improved visual outcomes following PRK if expanded LSCs are used to cover the cornea. The study will also compare the incidence of complications and characterize visual outcomes in patients treated with the new technique versus the control technique.

ELIGIBILITY:
Inclusion Criteria:

* Monocular corneal chemical injury or pterygium, or refractive error greater than +/- 2D
* Informed consent signed by patient or legal guardian

Exclusion Criteria:

* Patients with a history of corneal perforation or surgery
* Patients with other eye diseases
* Patients with a history of severe cardiovascular, liver, kidney, endocrine, and hematopoietic disease, diabetes, or immune deficiency disorders
* Pregnant or lactating women
* Patients who are participating in other clinical trials
* Patients with a history of mental illness who are unable to give informed consent or follow up according to the study protocol.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Composite measure of visual function in eyes treated for corneal ocular surface disease. | up to 1 year
  Slitlamp examination, in addition to measurement of visual acuity and intraocular pressure.
Composite measure of visual function in eyes after photo-refractive keratectomy (PRK) | up to 1 year

SECONDARY OUTCOMES:
Incidence of transparency of the cornea | up to 1 year
  Anterior segment photography and OCT as well as pentacam photography will be performed post treatment on day 1, week 1, week 2, month 1, month 3, month 6, and year 1, in order to assess transparency and curvature of the cornea.

OTHER OUTCOMES:
Postoperative complications | up to 1 year
  Slitlamp examination, anterior segment photography, anterior segment OCT, pentacam photography, in addition to measurement of visual acuity and intraocular pressure, will be performed post treatment on day 1, week 1, week 2, month 1, month 3, month 6, and year 1, in order to assess for any postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Kolli S, Ahmad S, Mudhar HS, Meeny A, Lako M, Figueiredo FC. Successful application of ex vivo expanded human autologous oral mucosal epithelium for the treatment of total bilateral limbal stem cell deficiency. Stem Cells. 2014 Aug;32(8):2135-46. doi: 10.1002/stem.1694. PMID 24590515
- [Background] Zakaria N, Possemiers T, Dhubhghaill SN, Leysen I, Rozema J, Koppen C, Timmermans JP, Berneman Z, Tassignon MJ. Results of a phase I/II clinical trial: standardized, non-xenogenic, cultivated limbal stem cell transplantation. J Transl Med. 2014 Mar 3;12:58. doi: 10.1186/1479-5876-12-58. PMID 24589151
- [Background] Vazirani J, Basu S, Kenia H, Ali MH, Kacham S, Mariappan I, Sangwan V. Unilateral partial limbal stem cell deficiency: contralateral versus ipsilateral autologous cultivated limbal epithelial transplantation. Am J Ophthalmol. 2014 Mar;157(3):584-90.e1-2. doi: 10.1016/j.ajo.2013.11.011. Epub 2013 Nov 19. PMID 24269851
- [Background] Wu Z, Zhou Q, Duan H, Wang X, Xiao J, Duan H, Li N, Li C, Wan P, Liu Y, Song Y, Zhou C, Huang Z, Wang Z. Reconstruction of auto-tissue-engineered lamellar cornea by dynamic culture for transplantation: a rabbit model. PLoS One. 2014 Apr 4;9(4):e93012. doi: 10.1371/journal.pone.0093012. eCollection 2014. PMID 24705327
- [Background] Konomi K, Satake Y, Shimmura S, Tsubota K, Shimazaki J. Long-term results of amniotic membrane transplantation for partial limbal deficiency. Cornea. 2013 Aug;32(8):1110-5. doi: 10.1097/ICO.0b013e31828d06d2. PMID 23615271
- [Background] Rama P, Matuska S, Paganoni G, Spinelli A, De Luca M, Pellegrini G. Limbal stem-cell therapy and long-term corneal regeneration. N Engl J Med. 2010 Jul 8;363(2):147-55. doi: 10.1056/NEJMoa0905955. Epub 2010 Jun 23. PMID 20573916
- [Background] Ouyang H, Xue Y, Lin Y, Zhang X, Xi L, Patel S, Cai H, Luo J, Zhang M, Zhang M, Yang Y, Li G, Li H, Jiang W, Yeh E, Lin J, Pei M, Zhu J, Cao G, Zhang L, Yu B, Chen S, Fu XD, Liu Y, Zhang K. WNT7A and PAX6 define corneal epithelium homeostasis and pathogenesis. Nature. 2014 Jul 17;511(7509):358-61. doi: 10.1038/nature13465. Epub 2014 Jul 2. PMID 25030175